CLINICAL TRIAL: NCT03090984
Title: Evaluation of Contact Phase Activation During Hemodialysis Using Different Dialysis Membranes: a Prospective Randomized Crossover Study
Brief Title: Evaluation of Contact Phase Activation During Hemodialysis
Acronym: c-phact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Karlien François, MD, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: UZB-NEF-2016-contactphase
Record Dates: First submitted 2017-02-10; First posted 2017-03-27 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; Coagulation activation
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PMMA (BKU) (Active Comparator): Patients included in the study will undergo 3 hemodialysis treatments. During the PMMA Arm, patient will be dialyzed using a BKU 1.6 (Toray) dialyzer. All study treatments will be standardized for dialysis access, priming procedure, blood and dialysate flows, anticoagulation therapy and duration of the hemodialysis session.
  During each study treatment, blood samples will be taken at specified time points (T0, T5, T15, T30, T90, T240) to assess overall coagulation activation (TAT, PF1+2, d-dimers), contact phase activation (kallikrein, fXIa, fXIIa), and activation of the extrinsic coagulation pathway (TF).
  Interventions: Device: PMMA (BKU)
- PS (Phylter) (Active Comparator): Patients included in the study will undergo 3 hemodialysis treatments. During the PS Arm, patient will be dialyzed using a Phylter 1.7 (Bellco) dialyzer. All study treatments will be standardized for dialysis access, priming procedure, blood and dialysate flows, anticoagulation therapy and duration of the hemodialysis session.
  Interventions: Device: PS (Phylter)
- AN69ST (Evodial) (Active Comparator): Patients included in the study will undergo 3 hemodialysis treatments. During the AN69ST Arm, patient will be dialyzed using a Evodial 1.6 (Gambro) dialyzer. All study treatments will be standardized for dialysis access, priming procedure, blood and dialysate flows, anticoagulation therapy and duration of the hemodialysis session.
  Interventions: Device: AN69ST (Evodial)

INTERVENTIONS:
Device: PMMA (BKU) — At serial time points before, during and after each study hemodialysis session using a BKU dialyzer, blood samples will be drawn for coagulation activation analyses.
  Arms: PMMA (BKU)
Device: PS (Phylter) — At serial time points before, during and after each study hemodialysis session using a Phylter dialyzer, blood samples will be drawn for coagulation activation
  Arms: PS (Phylter)
Device: AN69ST (Evodial) — At serial time points before, during and after each study hemodialysis session using an Evodial dialyzer, blood samples will be drawn for coagulation activation
  Arms: AN69ST (Evodial)

SUMMARY:
Every patient included in the study will undergo 3 standardised hemodialysis treatments, each using a different dialysis membrane (PMMA, PS, AN69ST). The order of the membranes used will be randomized.

During each conventional and standardised hemodialysis treatment, 6 blood samples will be taken at different time points (T0, T5, T15, T30, T90, T240) to evaluate coagulation activation (TAT, PF1+2, d-dimers, TF) and, more specifically, activation of the contact phase pathway of coagulation (kallikrein, fXIa, fXIIa).

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with hemodialysis since at least three months.
* Hemodialysis treatment schedule of 3 x 4 hours weekly.
* Arteriovenous fistula (AVF) use for vascular access.
* Treatment with oral acetylsalicylic acid 80 or 100mg q every day.
* ≥ 18 years of age.
* Patients able and agree to provide signed informed consent.

Exclusion Criteria:

* Use of vitamin K antagonists or novel oral anticoagulant therapy.
* Use of chronic heparin treatment, UFH or LMWH.
* Use of clopidogrel.
* Use of ACE-inhibitors.
* Known allergy against one of the dialysis membranes used during this study (PMMA: BKU®, Toray; PS: Phylter®, Bellco; AN69ST: Evodial®, Gambro).
* Known heparin-induced trombopenia type 2.
* Active infection and/or ongoing systemic antimicrobial treatment.
* Presence of central venous catheter, tunnelled or non-tunnelled and/or AV graft.
* Hospitalized patients.
* Planned surgery during study period.
* Mean Qb of <300ml/min during one of the last 3 dialysis sessions before inclusion.
* Vascular access dysfunction defined as (a) known AV access outflow tract stenosis, (b) planned vascular access intervention, (c) planned vascular access conversion.
* Planned conversion of dialysis modality during study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Change in contact phase activation induced by hemodialysis treatment, assessed by measurement of plasma kallikrein. | Blood samples are taken before hemodialysis treatment start and 5minutes (min), 15min, 30min, 90min and 240min after hemodialysis treatment start.
  ELISA testing for plasma kallikrein (pg/mL).
Change in contact phase activation induced by hemodialysis treatment, assessed by measurement of plasma fXIa. | Blood samples are taken before hemodialysis treatment start and 5min, 15min, 30min, 90min and 240min after hemodialysis treatment start.
  Chromogenic test for plasma fXIa (mIU/mL).
Change in contact phase activation induced by hemodialysis treatment, assessed by measurement of plasma fXIIa. | Blood samples are taken before hemodialysis treatment start and 5min, 15min, 30min, 90min and 240min after hemodialysis treatment start.
  ELISA testing for plasma fXIIa (pg/mL).

SECONDARY OUTCOMES:
Change in overall coagulation activation induced by hemodialysis treatment, assessed by measurement of plasma TAT. | Blood samples are taken before hemodialysis treatment start and 5min, 15min, 30min, 90min and 240min after hemodialysis treatment start.
  ELISA testing for plasma TAT (µg/L).
Change in overall coagulation activation induced by hemodialysis treatment, assessed by measurement of plasma PF1+2. | Blood samples are taken before hemodialysis treatment start and 5min, 15min, 30min, 90min and 240min after hemodialysis treatment start.
  ELISA testing for plasma PF1+2 (pmol/L).
Change in overall coagulation activation induced by hemodialysis treatment, assessed by measurement of plasma d-dimers. | Blood samples are taken before hemodialysis treatment start and 5min, 15min, 30min, 90min and 240min after hemodialysis treatment start.
  Immunoassay for plasma d-dimers (ng/mL)
Change in extrinsic coagulation activation during hemodialysis treatment assessed by measurement of plasma Tissue Factor | Blood samples are taken before hemodialysis treatment start and 5min, 15min, 30min, 90min and 240min after hemodialysis treatment start.
  ELISA testing for plasme Tissue Factor (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Karlien François, MD, Principal Investigator — UZ Brussel, Department of Nephrology
Locations (1):
- UZ Brussel, Jette, Belgium

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593